CLINICAL TRIAL: NCT03026049
Title: A Randomized Controlled Trial Comparing Venous Stenting With Conservative Treatment in Patients With Deep Venous Obstruction
Brief Title: Stent Versus Conservative Treatment in Patients With Deep Venous Obstruction
Acronym: STEVECO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: it was not possible to recruit the required amount of participants within a reseanable timefram.
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT DVO
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Deep-Venous Thrombosis; Deep Venous Stenting; Randomized Clinical Trial
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep venous stent (Active Comparator): Patients will receive deep venous stenting in the iliaco(femoral) region
  Interventions: Device: deep venous stenting
- conservative managment (No Intervention): Conservative management of complaints

INTERVENTIONS:
Device: deep venous stenting — Deep venous stent
  Arms: deep venous stent

SUMMARY:
Patients will be randomised between deep venous stenting or conservative management

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Meet criteria for PTS or
* Patients with May Thurner syndrome on additional imaging
* Life expectancy of more than one year
* Deep venous thrombosis > 1 year
* Signed informed consent

Exclusion Criteria:

* Previous intervention of central veins (inferior vena cava, iliac veins, common femoral vein) on the affected limb
* Known pregnancy
* Inability to answer Dutch QoL questionnaires or limited communication in Dutch (written and spoken)
* Contra-indication for prolonged anticoagulant treatment
* Recent, <1 year, deep venous thrombosis or pulmonary Embolism
* Known contrast allergy
* Known dialysis or renal insufficiency needing additional preparation for injection of contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life score | 12 months
  Quality of Life score

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht university medical center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829
- [Derived] Shekarchian S, Van Laanen J, Esmaeil Barbati M, Vleugels MJ, Nelemans P, Razavi MK, Mees B, Jacobs MJ, Jalaie H. Editor's Choice - Quality of Life after Stenting for Iliofemoral Venous Obstruction: A Randomised Controlled Trial with One Year Follow Up. Eur J Vasc Endovasc Surg. 2023 Nov;66(5):678-685. doi: 10.1016/j.ejvs.2023.07.044. Epub 2023 Jul 28. PMID 37517579
- [Derived] van Vuuren TM, van Laanen JHH, de Geus M, Nelemans PJ, de Graaf R, Wittens CHA. A randomised controlled trial comparing venous stenting with conservative treatment in patients with deep venous obstruction: research protocol. BMJ Open. 2017 Sep 11;7(9):e017233. doi: 10.1136/bmjopen-2017-017233. PMID 28893753